# STATISTICAL ANALYSIS PLAN

| Document title | Statistical analysis plan of trial as per protocol SG-2/1215 |
|---|---|
| Version No. | Final, 1.2 |

| Treatment groups | Seroguard, 1.5 and 2.4 mL/kg; Placebo |
|---|---|
| Protocol No. | SG-2/1215 |
| Protocol title | Phase II multi-center, randomized, double-blind, placebo-controlled efficacy and dose ranging trial of the drug product Seroguard, solution (JSC Pharmasyntez, Russia) used for the prevention of pelvic adhesions. |
| Sponsor | JSC Pharmasyntez, Russia |
| CRO | CROMOS PHARMA LLC |
| Data processing center | KEYSTAT LLC |

| Document version control | | |
|---|---|---|
| Version | Modification date | Modification cause |
| Preliminary version 1.0 | April 14, 2017 | Primary version |
| Preliminary version 1.1 | April 17, 2017 | Amendment in the description of MRI efficacy variables |
| Preliminary version 1.2 | April 19, 2017 | Amendments according to the Sponsor comments |
| Final 1.2 | April 24, 2017 | Document approved |

| D. Khamtsov President, KEYSTAT LLC | | «» 2017 |
|---|---|---|
| I. Murashko Project manager, CROMOS PHARMA LLC | /signed/ | «28» April 2017 |
| M.G. Shurygin R & D Director, JSC Pharmasyntez | /signed/ | «02» <b>M</b> ay 2017 |

By receiving the document you agree that it is a confidential intellectual property of JSC Pharmasyntez. You shall never directly or indirectly publish, distribute or otherwise disclose content of the document and make any part of it available to a third party. The document must be used solely for the purpose it was given to you. Information can be disclosed only subject to the prior written authorization of JSC Pharmasyntez or to representatives of authorized government bodies or pursuant to an order from a court. JSC Pharmasyntez shall be immediately notified about any disclosure of information contained in the document (authorized or otherwise).

# **TABLE OF CONTENTS**

| 1. | INTR | ODUCTION | 6 |
|---|---|---|---|
| 2. | LIST | OF ABBREVIATIONS | 7 |
| 3. | STUE | DY DESIGN | 9 |
| | 3.1 | Randomization | 9 |
| | 3.2 | Blinding | 10 |
| | 3.3 | Study drugs | 11 |
| 4. | STUE | DY OBJECTIVES | 13 |
| | 4.1 | Primary objectives | 13 |
| | 4.2 | Secondary objectives: | 13 |
| 5. | DETE | ERMINATION OF THE SAMPLE SIZE | 14 |
| 6. | MISS | ING DATA SUBSTITUTION | 16 |
| 7. | ANAL | YSIS POPULATIONS | 16 |
| | 7.1 | Efficacy analysis set | 16 |
| | | 7.1.1 Intent-to-treat (ITT) | 16 |
| | 7.0 | 7.1.2 Per-protocol (PP) | 16 |
| _ | 7.2 | Safety population | 17 |
| 8. | | ENT POPULATION | 17 |
| | 8.1 | Patient disposition | 17 |
| ^ | 8.2 | Demographic and other baseline characteristics | 17 |
| 9. | | CACY AND SAFETY VARIABLES | 18 |
| | 9.1 | Primary efficacy variable | 18 |
| | 9.2 | Secondary efficacy variables | 18 |
| 40 | 9.3 | Safety variables | 18 |
| 10. | | CACY ANALYSIS | 19 |
| | 10.1 | Primary efficacy variable | 19 |
| 44 | 10.2 | Secondary efficacy variables | 20 |
| 11. | | TY ANALYSIS | 20 |
| | 11.1 | Assessment of adverse events and serious adverse events | 21 |
| | 11.2 | Laboratory data evaluation | 22 |
| | 11.3 | Concomitant therapy | 22 |
| | 11.4<br>11.5 | Abdominal ultrasound 12-lead ECG | 22 |
| | 11.6 | | 22 |
| | | Vital Signs Assessment | 23 |
| | 11.7<br>11.8 | Physical examination Pastaparative wound assessment | 23<br>23 |
| 10 | | Postoperative wound assessment RIM ANALYSIS | 23 |
| 12. | | | |
| 13.<br>14. | | ERAL PROVISIONS<br>E TEMPLATES | 23 |
| 1 <del>4</del> . | 14.1 | | 24<br>24 |
| | 14.1<br>14.2 | Demographic and Other Baseline Characteristics Efficacy Analysis | 29 |
| | 14.4 | 14.2.1 Primary efficacy variable | 29<br>29 |

| i-2/1215 Sta | tistical Analysis Plan | Final version 1.2 |
|--------------|-------------------------------------|-------------------|
| | 14.2.2 Secondary efficacy variables | 29 |
| 14.3 | Safety Analysis | 34 |

# List of tables

| TABLE 3.1 SCHEDULE OF VISITS AND STUDY PROCEDURES | 12 |
|---|---|
| TABLE 14.1 PATIENT DISPOSITION | 24 |
| TABLE 14.2 REASONS OF PATIENTS EXCLUSION FROM THE PP POPULATION | 24 |
| TABLE 14.3 REASONS OF PATIENTS EXCLUSION FROM THE ITT POPULATION | 24 |
| TABLE 14.4 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS. SCREENING. ITT POPULATION. N | |
| = XX | 24 |
| TABLE 14.5 DATA ON DISEASE. SCREENING. ITT POPULATION. N = XX | 25 |
| TABLE 14.6 PREVIOUS DISEASES. ITT POPULATION. SCREENING. N = XX | 27 |
| TABLE 14.7 CONCURRENT DISEASES. ITT POPULATION. SCREENING. N = XX | 27 |
| TABLE 14.8 PRIOR THERAPY. SCREENING. ITT POPULATION. N = XX | 27 |
| TABLE 14.9 PHYSICAL EXAMINATION. ITT POPULATION. SCREENING. N = XX | 27 |
| TABLE 14.10 HIV, RW, HBV AND HCV TEST RESULTS. ITT POPULATION. N = XX | 28 |
| TABLE 14.11 PREGNANCY TEST. SCREENING. ITT POPULATION. N = XX | 28 |
| TABLE 14.12 12-LEAD ECG. SCREENING. ITT POPULATION. N = XX | 28 |
| TABLE 14.13 VITAL SIGNS. ITT POPULATION. SCREENING. N = XX | 28 |
| TABLE 14.14 TREATMENT SUCCESS. DECREASE IN THE NUMBER OF ADHESIONS. ITT POPULATION. N = | |
| XX | 29 |
| TABLE 14.15 TREATMENT SUCCESS. DECREASE IN THE NUMBER OF ADHESIONS. PP POPULATION. N = | |
| XX | 29 |
| TABLE 14.16 ASSESSMENT OF ADHESION SEVERITY BY PAI (PELVIC ADHESIONS INDEX) | 29 |
| TABLE 14.17 NUMBER OF HYPERECHOIC LINEAR LESIONS POST SURGERY AS BASED ON TRANSVAGINAL | |
| ULTRASOUND RESULTS. ITT POPULATION. N = XX | 30 |
| TABLE 14.18 LIMITED MOBILITY OF PELVIC ORGANS POST SURGERY. ITT POPULATION. N = XX | 31 |
| TABLE 14.19 ABSENCE OF PELVIC ADHESIVE DISEASE SIGNS. ITT POPULATION. N = XX | 32 |
| TABLE 14.20 THICKNESS OF ADHESIONS. ITT POPULATION. N = XX | 33 |
| TABLE 14.21 EXTENT OF THE ADHESION PROCESS IN THE PELVIC CAVITY. | 34 |
| TABLE 14.22 12-LEAD ECG DURING THE STUDY. SAFETY POPULATION. N = XX | 34 |
| TABLE 14.23 12-LEAD ECG DURING THE STUDY. ABSOLUTE VALUES. SAFETY POPULATION. N = XX | 35 |
| TABLE 14.24 ABDOMINAL ULTRASOUND DURING THE STUDY. SAFETY POPULATION. N = XX | 35 |
| TABLE 14.25 PHYSICAL EXAMINATION. SAFETY POPULATION. N = XX | 36 |
| TABLE 14.26 LOCAL STATUS ASSESSMENT. SAFETY POPULATION. N = XX | 37 |
| TABLE 14.27 PREGNANCY TEST. SAFETY POPULATION. N = XX | 38 |
| TABLE 14.28 CONCOMITANT THERAPY DURING THE STUDY. SAFETY POPULATION. N = XX | 38 |
| TABLE 14.29 VITAL SIGNS. SAFETY POPULATION. N = XX | 39 |
| TABLE 14.30 LABORATORY DATA EVALUATION. COAGULOGRAM. SAFETY POPULATION. N = XX | 39 |
| TABLE 14.31 LABORATORY DATA EVALUATION. COAGULOGRAM. ABNORMAL FINDINGS ONLY. | 39 |
| TABLE 14.32 LABORATORY DATA EVALUATION. COMPLETE BLOOD COUNT. SAFETY POPULATION. N = XX | 40 |
| TABLE 14.33 LABORATORY DATA EVALUATION. COMPLETE BLOOD COUNT. ABNORMAL FINDINGS ONLY. | 44 |
| SAFETY POPULATION. N = XX TABLE 14 24 LABORATORY DATA EVALUATION, BLOOD BLOCKLENICTRY, CAFETY POPULATION, N XX | 41 |
| TABLE 14.34 LABORATORY DATA EVALUATION. BLOOD BIOCHEMISTRY. SAFETY POPULATION. N = XX | 41 |
| TABLE 14.35 LABORATORY DATA EVALUATION. BLOOD BIOCHEMISTRY. ABNORMAL FINDINGS ONLY. | 44 |
| SAFETY POPULATION. N = XX TABLE 14 26 LABORATORY DATA EVALUATION LUBINALIZES CAFETY POPULATION N. XXX | 41 |
| TABLE 14.36 LABORATORY DATA EVALUATION. URINALYSIS. SAFETY POPULATION. N = XX | 41 |
| TABLE 14.37 LABORATORY DATA EVALUATION. URINALYSIS. ABNORMAL FINDINGS ONLY. SAFETY POPULATION. N = XX | 41 |
| TABLE 14.38 BRIEF SUMMARY OF ADVERSE EVENTS. SAFETY POPULATION. N = XX | 41<br>42 |
| TABLE 14.39 ADVERSE EVENTS. SAFETY POPULATION. N = XX | 42 |
| TABLE 14.40 SERIOUS ADVERSE EVENTS. SAFETY POPULATION. N = XX | 42 |
| TABLE 14.41 ADVERSE EVENTS BY THE DEGREE OF SEVERITY. SAFETY POPULATION. N = XX | 43<br>43 |
| TABLE 14.42 SERIOUS ADVERSE EVENTS BY THE DEGREE OF SEVERITY. SAFETY POPULATION. N = XX | 43<br>44 |
| TABLE 14.43 ADVERSE EVENTS AND THEIR RELATION TO THE STUDY DRUG. SAFETY POPULATION. N = XX | 44 |
| XX | 44 |
| TABLE 14.44 SERIOUS ADVERSE EVENTS AND THEIR RELATION TO THE STUDY DRUG. SAFETY | 44 |
| POPULATION. N = XX | 45 |
| TABLE 14 45 LABORATORY DATA EVALUATION COMPLETE BLOOD COUNT ABSOLUTE VALUES SAFETY | 73 |

| SG-2/1215 Statistical Analysis Plan | Final version 1.2 |
|---|---|
| POPULATION. N = XX | 45 |
| TABLE 14.46 LABORATORY DATA EVALUATION. BLOOD BIOCHEMISTRY. ABSOLUTE VALUES. SAFET | Υ |
| POPULATION. N = XX | 46 |
| TABLE 14.47 LABORATORY DATA EVALUATION. URINALYSIS. ABSOLUTE VALUES. SAFETY POPULAT | ION. N |
| = XX | 46 |
| TABLE 14.48 LABORATORY DATA EVALUATION. COAGULOGRAM. ABSOLUTE VALUES. SAFETY | |
| POPULATION. N = XX | 46 |

# 1. INTRODUCTION

This document describes the planned statistical analysis of clinical trial data (JSC Pharmasyntez) as per protocol SG- 2/1215: Phase II multi-center randomized double-blind placebo-controlled efficacy and dose ranging trial of the drug product Seroguard, solution (JSC Pharmasyntez, Russia) used for the prevention of pelvic adhesions.

# 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| AE | Adverse event |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| APTT | Activated partial thromboplastin time |
| AR | Adverse reaction |
| ASA | American Association of Anaesthetists |
| AST | Aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical classification system |
| BADS | Biologically Active Dietary Supplements |
| ВМІ | Body Mass Index = Weight/Height (cm) <sup>2</sup> |
| BP | Blood pressure |
| CI | Confidence interval |
| COX | Cyclooxygenase |
| CRF | Case Report Form |
| CRO | Contract research organization |
| DBP | Diastolic blood pressure |
| EC | Ethics Committee |
| ECG | Electrocardiogram |
| ESR | Erythrocyte sedimentation rate |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GGT | Gamma-glutamyl transpeptidase |
| HIV | Human immunodeficiency virus |
| HR | Heart rate |
| ICD | International classification of diseases |
| ICH | The International Conference on Harmonization of Technical |
| ICH | Requirements for Registration of Pharmaceuticals for Human Use |
| ICH GCP | International Conference on Harmonization Good Clinical Practice |
| ICH GCF | Guidelines |
| INN | International nonproprietary name |
| INR | International normalized ratio |
| ІТТ | Intent-to-treat, or population comprising all patients included in the |
| | trial |
| LEC | Local ethics committee |
| LLN | Lower limit of normal |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mm Hg | millimeter of mercury |
| NEC | National ethics committee |
| PAI | Pelvic Adhesions Index |
| PATE | Pulmonary artery thromboembolia |
| PP | Per protocol, or population of patients who completed the trial as |
| | per protocol |
| RNA | Ribonucleic acid |
| RR | Respiratory rate |
| SAE | Serious adverse event |
| SAR | Serious adverse reaction |
| SBP | Systolic blood pressure |
| SOP | Standard operating procedure |
| TESS | Treatment Emergency Sign and Symptom |

| Abbreviation | Definition |
|--------------|---------------------------|
| ULN | Upper limit of normal |
| WHO | World Health Organization |
| WMO | World Medical Association |

#### 3. STUDY DESIGN

A multi-center, randomized, double-blind, placebo-controlled efficacy and dose ranging clinical trial of the drug product Seroguard, solution (JSC Pharmasyntez, Russia) used for the prevention of pelvic adhesions will be performed.

After a female patient successfully completes screening procedures she will undergo a planned laparoscopic operation. All patients will be randomized into treatment groups at the surgery date with the help of on-line IWRS system (Interactive Web Response System). The test drug or placebo are administered at the final stage of the surgery. After the surgery, a patient will stay in hospital for a 6-day observation period. At day 7, unless clinically contraindicated, a patient can be discharged from hospital and will be further observed on an outpatient basis. The observation period duration is 4 weeks up to day 28 of the study. Then a final evaluation of the treatment efficacy is carried out at the repeated MRI of the abdomen and pelvis.

Trial procedures for evaluation of safety and efficacy of the test drug and placebo will be the same in all treatment groups:

- 1) group of placebo, 1.5 mL/kg up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases;
- 2) group of placebo, 2.4 mL/kg up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases;
- 3) group of Seroguard, 1.5 mL/kg up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases;
- 4) group of Seroguard, 2.4 mL/kg up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases.



Figure 3.1 Study Design Flowchart

# 3.1 RANDOMIZATION

After female patients sign the informed consent form to participate in the study and it is

confirmed that they meet the inclusion criteria and do not have the non-inclusion criteria they will be allocated into treatment groups by means of a centralized block randomization in a 1:1:11 ratio without stratification by the study centre via on-line IWRS system (Interactive Web Response System). A study subject will be assigned a randomization ID in the order of access to the IWRS system. Randomization IDs corresponding to the test drug or placebo administration will be randomly assigned to the equal number of patients.

- 1. Placebo, 1.5 mL/kg group up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases.
- 2. Placebo, 2.4 mL/kg group up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases.
- 3. Seroguard, 1.5 mL/kg group up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases.
- 4. Seroguard, 2.4 mL/kg group up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases.

A block generation of the randomization sequence will be used to generate a randomization list. The randomization list will be generated by a statistics software using a random number generator at the stage of preparation to the study.

It is only a patient's randomization ID that will be recorded in the CRF with no specification of the administered drug.

Investigators will have an online training on using the IWRS system.

A register of screened and randomized patients will be maintained for all study centers. The register form is provided in the Study Center File. It should be regularly filled in by investigators entering all the data required.

For patients to be identified in case of an insured event, each of them will be assigned a unique identification code created by the following scheme:

- Study authorization number;
- Date the study authorization was issued in the DD MM YYYY format;
- Medical organization number specified in the authorization;
- Patient's initials (first letters of her surname, name and patronymic);
- Patient's birthday in the DD MM YYYY format;
- Patient's unique number (can consist of digits and/or letters).

| Stud<br>authoriz<br>numb | zation | Date | study<br>was i<br>O MN | issue | ed | n org | numl<br>ecific<br>the | ation<br>per<br>ed in | i<br>(fin<br>su<br>na | of he<br>irnan<br>ime a | ls<br>ters<br>r<br>ne, | Pati<br>(DD | ( | tient<br>cons | ist o | r |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

#### 3.2 BLINDING

The present trial is designed as a double-blind, placebo-controlled study. In order to provide the maximum objective evaluation of the primary endpoint neither a medical

Investigator, nor patients will have access to the treatment assignment code.

Blinding is performed in such a way that disclosing a randomization code of a certain subject excludes a disclosure of the code in general (i.e. the randomization code has no indication of the treatment group).

In order to ensure the double blind design of the study, an unblinded pharmacist will be included in a study team of the investigation site. The unblinded pharmacist will distribute a study drug for a particular patient by using the IRWS system, calculate the volume of the drug to be administered (mL) to each patient according to the treatment group and data on the patient's weight, and prepare the drug immediately prior to its administration to the patient in accordance with the "Study drug preparation instructions for unblinded study team members" (provided to study centers as a separate document).

An unblinded pharmacist of the study team must not inform a site representative or other blinded team members, or Sponsor representative/blinded CRO representative on the treatment group (except for cases when unblinding is necessary to make a decision on the further strategy of a patient treatment). A fact of unblinding as well as reasons of an inquiry for information unblinding are to be recorded in the patient's primary documentation in detail.

#### 3.3 STUDY DRUGS

- 1. Placebo, 1.5 mL/kg group up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases.
- 2. Placebo, 2.4 mL/kg group up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases.
- 3. Seroguard, 1.5 mL/kg group up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases.
- 4. Seroguard, 2.4 mL/kg group up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases.

Table 3.1 Schedule of Visits and Study Procedures

| | | Concadie of V | | I. | | |
|---|---|---|---|---|---|---|
| | Screening | Surgery | Obser | vation | | |
| Procedures | Visit 0 | Visit 1 | Visit 2 | Visit 3 | Unscheduled visit <sup>1</sup> | Early termination visit |
| Troccuares | Day -15<br>to -1 | Day 0 | Day 6±1 | Day 30±4 | Clisticuated visit | Larry termination visit |
| Informed consent | + | | | | | |
| Evaluation of the inclusion, non-inclusion criteria | + | + | | | | |
| Evaluation of the withdrawal criteria | | | + | | + | |
| Collection of medical and pharmacotherapeutic analysis data | + | | | | | |
| Collection of demographic and anthropometric data | + | | | | | |
| Physical examination | + | + | + | + | + | + |
| Local status assessment | | + | + | + | + | +2 |
| Measurement of vital signs <sup>3</sup> | + | + | + | + | + | + |
| HIV, RW, HBV and HCV blood test | + | | | | | |
| Pregnancy test | + | | | + | | + |
| Randomization | | + | | | | |
| Complete blood count | + | | + | + | + | + |
| Blood biochemistry | + | | + | + | + | + |
| Coagulogram | + | | | + | | + |
| Urinalysis | + | | + | + | + | + |
| Abdominal /pelvic MRI | + | | | + | | + |
| Abdominal ultrasound | + | | + | | | + |
| Pelvic ultrasound | + | | | + | | + |
| Gynecological examination and colposcopy | + | | | | | |
| Cervical cytology by Pap smears | + | | | | | |
| Smear microscopy | + | | | | | |
| Hysterosalpingography <sup>4</sup> | + | | | | | |
| 12-lead ECG | + | | + | + | + | + |
| Concomitant therapy evaluation | | + | + | + | + | + |
| Administration of the test drug/placebo | | + | | | | |
| Detection of ARs | + | + | + | + | + | + |

<sup>&</sup>lt;sup>1</sup> Any additional study procedure can be performed if indicated, at the discretion of the Principal Investigator

<sup>&</sup>lt;sup>2</sup> If applicable

<sup>&</sup>lt;sup>3</sup> Blood pressure, heart rate at the radial artery, respiration rate, body temperature will be measured.

<sup>&</sup>lt;sup>4</sup> Performed at the discretion of a doctor for women diagnosed with infertility who are enrolled in the study.

#### 4. STUDY OBJECTIVES

The trial is aimed at evaluating efficacy of Seroguard solution used for the prevention of pelvic adhesions.

#### 4.1 PRIMARY OBJECTIVES

To compare the efficacy of Seroguard solution administered at the dose of 1.5 or 2.4 mL/kg and the placebo (1.5 or 2.4 mL/kg of 0.9 % sodium chloride solution) in terms of presence, severity and extent of adhesions after laparoscopic treatment of pelvic adhesions in female patients.

To evaluate the safety profile of Seroguard solution administered at the dose of 1.5 or 2.4 mL/kg as compared to the placebo (1.5 or 2.4 mL/kg of 0.9 % sodium chloride solution) after laparoscopic treatment of pelvic adhesions.

#### 4.2 SECONDARY OBJECTIVES:

- 1. to determine a change in the number of pelvic adhesions as based on postsurgery MRI data in comparison to pre-surgery MRI data;
- 2. to determine a change in thickness of pelvic adhesions as based on postsurgery MRI data in comparison to pre-surgery MRI data;
- 3. to determine a frequency of detecting limited mobility of pelvic organs post surgery (as based on transvaginal ultrasound results);
- 4. to determine a frequency of hyperechoic linear lesion detection post surgery as based on transvaginal ultrasound results;
- 5. to determine a change in the frequency of detecting pelvic organ limited mobility in comparison to the baseline (absolute change and percentage from the baseline);
- 6. to determine a change in frequency of hyperechoic linear lesion detection as based on results of a repeated transvaginal ultrasound in comparison to the baseline:
- to determine a frequency of detecting no ultrasound signs of pelvic adhesive disease post surgery (defined as no limited mobility of pelvic organs and no hyperechoic linear lesions);
- 8. to determine a number of adhesions at the surgery;
- 9. to determine a number of dense adhesions at the surgery;
- 10. to determine a percentage of patients with any adverse reactions;
- 11. to determine a percentage of patients with any serious adverse reactions;
- 12. to determine a percentage of patients with adverse reactions "definitely", "probably" or "possibly" related to the test drug or the placebo;
- 13. to determine a percentage of female patients with serious adverse reactions "definitely", "probably" or "possibly" related to the test drug or the placebo;
- 14. to determine a percentage of patients with mild adverse reactions;
- 15. to determine a percentage of patients with moderate adverse reactions;
- 16. to determine a percentage of patients with severe adverse reactions;

- 17. to determine a percentage of patients with clinically significant changes in physical examination results:
- 18. to determine a percentage of patients with clinically significant changes in vital signs;
- 19. to determine a percentage of patients with clinically significant changes in ECG results:
- 20. to determine a percentage of patients with clinically significant changes in laboratory test results.

## 5. DETERMINATION OF THE SAMPLE SIZE<sup>1</sup>

In the studies of Adept® (Innoventica plc) that is the closest drug to the test one by its mechanism of action (U.S. Food and Drug Administration, 2006), a primary endpoint defined as a decrease in the number of adhesions by 3 or more (in patients with 10 or less adhesions at the baseline) or by 30% and more (in patients with >10 adhesions at the baseline) at the second look diagnostic laparoscopy was used and it was achieved in 45 %.

As soon as performance of a second look laparoscopy in the present trial is ethically unacceptable, MRI will be used for the purpose of primary endpoint evaluation. According to the publication (Ghonge & Ghonge, 2014) MRI results strongly correlate to those of a diagnostic laparoscopy (including both pre- and post-surgery examinations at second look laparoscopies). The only exceptions are the thinnest adhesions that cannot be visualized by MRI but for this purpose high field MRI can be performed. Hence, MRI allows to visualize adhesions both in terms of their quality and quantity and to obtain data with the same degree of detalization as during pre- and post-surgery laparoscopic examination.

Thus, the size will be calculated on the basis of efficacy of similar drugs studied on the laparoscopy data basis, however, in the present trial MRI control will be used first and for most due to ethical considerations and due to a strong correlation between MRI and laparoscopy data.

According to the above Adept® studies (U.S. Food and Drug Administration, 2006), the primary endpoint effectiveness (clinical success determined as a decrease in the number of adhesions at the second look diagnostic laparoscopy by 3 and more (in patients with 10 or less adhesions at the baseline) or by 30% and more (in patients with > 10 adhesions at the baseline)) is 45%. According to the literature review and meta-analysis (Ahmad, et al., 2014), clinical efficacy in the control group (placebo) is achieved in no more than 10% cases.

Using these baseline data, the following assumptions are made (as per the method specified in (U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), Center for Biologics Evaluation and Research (CBER), 2010)):

1. The study will be conducted as a superiority trial, i.e. at least one dosage of Seroguard is to be more efficient than the placebo with the superiority margin of 5% and more (definition of the endpoint and superiority margin given in the main pivotal of Adept<sup>®</sup> is used). Each dosage of the test drug will be compared with the placebo separately. Comparison of the two dosages of the test drug by their

\_

<sup>&</sup>lt;sup>1</sup> Cited by the Study protocol

efficacy is not planned and it will be studied in phase III clinical trials.

- 2. Expected rates of achieving the primary endpoint in the different dosage groups will be considered as initially equal.
- 3. First type error ( $\alpha$ ) for the superiority hypothesis is 5% (0.05).
- 4. Second type error (β) is set at 20 % (0.2) which corresponds to 80% power.
- 5. Expected withdrawal rate at screening is 15% and after randomization 10%.

Null and alternative hypotheses for the *superiority testing* are as follows:

The null hypothesis (H<sub>0</sub>) holds that the difference in the rate of the primary endpoint achievement between one of the Seroguard dosages and the placebo will not exceed 5% in favor of the drug

$$H_0: p_1 - p_0 \le 0.05$$

The alternative hypothesis (H<sub>A</sub>) holds that the difference in the rate of the primary endpoint achievement between one of the Seroguard dosages and the placebo will exceed 5% in favor of the drug

$$H_A$$
:  $p_1 - p_0 > 0.05$ 

where p<sub>0</sub> and p<sub>1</sub> are the rates of the primary endpoint achievement in the groups of the placebo and Seroguard (at any dosage), respectively.

In this case for the purpose of the sample size calculation in each group the formula given in: Chow S, Shao J, Wang H. Sample Size Calculations in Clinical Research. 2nd ed.: Chapman&Hall / CRC Biostatistics Series; 2008, is employed:

$$n = (p_1 \times (1 - p_0) + p_0 \times (1 - p_0)) \times \left(\frac{z_{1-\alpha} + z_{1-\beta}}{p_1 - p_0 - \delta}\right)^2$$

where

n is the size of a group;

z is the value of the normal distribution function at the given  $\alpha$  and  $\beta$  levels;

 $\delta$  is the superiority margin – 5%;

p<sub>1</sub> is the expected percentage in the test drug group (at any dosage) – 45%;

 $p_0$  is the expected percentage in the placebo group -5%.

By inserting the above data in the formula a minimum of patients in the placebo group without consideration of their withdrawal rate is calculated: 24 completed cases which corresponds to 26 randomized and 30 screened patients.

Thus, the total number of patients to be enrolled in the study is:

- 1. Placebo, 1.5 mL/kg group up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases;
- 2. Placebo, 2.4 mL/kg group up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases;
- 3. Seroguard, 1.5 mL/kg group up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases;
- 4. Seroguard, 2.4 mL/kg group up to 30 screened patients which corresponds to 26 randomizations and 24 completed cases.

Thus, 120 female patients are to be screened and at least 104 are to be randomized.

# 6. MISSING DATA SUBSTITUTION

Substitution of missing data will be performed only in the adverse event (AE) analysis.

In order to determine whether a certain AE is a study event (TESS – Treatment Emergency Sign and Symptom) missing dates of AE starting will be substituted by using the following algorithm:

AEs with a missing starting date will included in the analysis.

If an AE starting date is incomplete the following rules should be applied:

| Day | Month | Year | AE is included in the analysis if |
|---|---|---|---|
| Missing | Present | Present | the month and year is ≥ the date of the first drug dose administration (month and year). |
| Missing | Missing | Present | the year is ≥ the year of the first drug dose administration |
| Present | Missing | Missing | The worst variant. Included |
| Present | Present | Missing | The worst variant. Included |
| Present | Missing | Present | the year is ≥ the year of the first drug dose administration |
| Missing | Present | Missing | the month is ≥ the month of the first drug dose administration (it is assumed that the year is 2017). |

If the relationship with the drug is missing the given AE is classified as "related".

#### 7. ANALYSIS POPULATIONS

A patient's classification into a particular analysis population will be approved by the study Sponsor prior to the statistical analysis.

#### 7.1 EFFICACY ANALYSIS SET

#### 7.1.1 Intent-to-treat (ITT)

The ITT set also known as the full analysis set includes all randomized patients exposed to the drug regardless of their compliance with the protocol throughout the study. This is the main analysis set and it will be used for evaluation of all planned parameters.

A patient's classification into the ITT population will be made prior to the analysis and is a subject to the Sponsor approval.

#### 7.1.2 Per-protocol (PP)

In addition to analysis as per ITT all planned parameters will be also analyzed with the use of the patients data selected by the principle of a patient's compliance with the protocol (PP). The given population won't be analyzed, if it is more than 90% and less than 50% of the ITT population. A patient's data are to be excluded from the PP data set in the following cases:

- the inclusion and non-inclusion criteria are significantly violated;
- forbidden concomitant therapy is used;
- any other major violation of the protocol considered as significantly violating the primary efficacy evaluation in the given study subject.

A patient's classification into the PP population will be made prior to the analysis and is a subject to the Sponsor approval.

#### 7.2 SAFETY POPULATION

The data set for the safety evaluation analysis is identical to the ITT data set. But, in contrast to the intent-to-treat population, all subjects data are analyzed depending on the actual treatment received (if it different from the one that was assigned via randomization). All safety analyses will be based on the safety analysis data set.

#### 8. PATIENT POPULATION

The ITT population is considered the primary analysis population. An additional analysis of the primary efficacy endpoint will also be performed in the PP population to confirm the results obtained.

The groups of placebo at different dosages are merged into one to be compared with the groups of Seroguard 1.5 mL/kg and 2.4 mL/kg.

#### 8.1 PATIENT DISPOSITION

The number of screened patients, that of randomized (included in the study) patients, number of subjects in the populations under analysis and of subjects who completed the study will be presented by treatment groups.

#### 8.2 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic characteristics will be described by treatment groups in the ITT population (primary population for the efficacy analysis):

- age,
- race,
- sex (female only),
- height,
- body weight,
- BMI.
- physical examination,
- vital signs,
- pregnancy test,
- prior therapy,
- previous diseases,
- concomitant diseases,
- underlying disease information,
- HIV, RW, HBV and HCV blood test results,
- gynecological examination and colposcopy,
- smear cytology and microscopy,
- hysterosalpingography,
- 12-lead ECG (abnormalities only).

The treatment groups will be compared by the following demographic and baseline characteristics:

- age,
- BMI.
- symptoms and parameters of the disease,

physical examination data.

Treatment groups will be compared by using a mixed linear model where a study center is a random factor. The hypothesis that the three groups are equal is tested.

The intergroup comparison of physical examination data and ECG abnormalities will be carried out by using Fisher's exact test.

The treatment group comparison by parameters of the disease will be performed with the use of either Fisher's exact test (for nominal data) or a mixed linear model (ANOVA) (for continuous data). All tests are given in table templates.

Concurrent and previous diseases will be coded by the MedDRA dictionary and presented in groups by the System Organ Class (SOC) and Preferred Terms (PT).

The comparison of treatment groups by the below parameters won't be carried out:

- vital signs,
- pregnancy test,
- previous diseases,
- concomitant diseases.
- HIV, RW, HBV and HCV blood test results.

## 9. EFFICACY AND SAFETY VARIABLES

#### 9.1 PRIMARY EFFICACY VARIABLE

Achieving clinical efficacy of the drug determined as:

 frequency of reduction of the adhesions number at the repeated MRI by 3 or more (in patients with 10 and less adhesions at the baseline) or by 30% and more (in patients with >10 adhesions at the baseline) in comparison to baseline MRI data.

## 9.2 SECONDARY EFFICACY VARIABLES

- 1. change in the thickness of pelvic adhesions by a repeated MRI in comparison to baseline MRI data;
- 2. frequency of detecting pelvic organs limited mobility post surgery (based on transvaginal ultrasound results) on Day 30±4 after surgery;
- 3. frequency of detection of hyperechoic linear lesions post surgery as based on transvaginal ultrasound results;
- 4. change in the frequency of detecting pelvic organs limited mobility in comparison to the baseline (absolute change and percentage from the baseline);
- 5. change in the frequency of hyperechoic linear lesion detection as based on results of a repeated transvaginal ultrasound in comparison to the baseline;
- 6. frequency of detecting no ultrasound signs of pelvic adhesive disease post surgery (defined as no limited mobility of pelvic organs and no hyperechoic linear lesions).

#### 9.3 SAFETY VARIABLES

Vital signs (body temperature, blood pressure, HR, RR)

- Laboratory test results:
  - blood biochemistry total protein, glucose, ALT, AST, total bilirubin, alkaline phosphatase, amylase, creatinine;
  - complete blood count RBC, WBC, platelet count, haemoglobin, hematocrit, WBC differential, ESR;
  - coagulogram coagulation time, international normalized ratio (INR), thrombin time, activated partial thromboplastin time (APTT);
  - o urinalysis color, transparency, pH, specific gravity, protein, glucose, WBC, RBC, bacteria, casts, salts.
- ECG data heart rate [HR]; PR, QRS, QT intervals and calculated QTc interval.
- Ultrasound data
- Incidence of adverse reactions
- Incidence of serious adverse reactions
- Incidence of unexpected adverse reactions
- Incidence of adverse and serious adverse reactions resulting in treatment discontinuation/withdrawal from the study

#### 10. EFFICACY ANALYSIS

If treatment groups show a statistically significant difference this issue will be discussed separately with the Sponsor. In such case it may be necessary to consider a possibility of building a logistic model and deriving required CI limits from it.

#### 10.1 PRIMARY EFFICACY VARIABLE

#### The analysis is performed both in the ITT and PP populations.

Treatment success is defined as:

 frequency of reduction of the adhesions number at the repeated MRI by 3 or more (in patients with 10 and less adhesions at the baseline) or by 30% and more (in patients with >10 adhesions at the baseline) in comparison to baseline MRI data.

Null hypothesis (H0) is worded in the following way: the test drug (Seroguard at the dose of XX) is superior to the reference drug (placebo) by the primary endpoint.

The hypothesis testing is:

Null hypothesis 
$$H_0$$
:  $p_T - p_R \le d$ 

Alternative hypothesis 
$$H_1$$
:  $p_T - p_R > d$ 

where  $p_T$  is the treatment success ratio in the group of the test drug Seroguard at a certain dose (T, test);

 $p_R$  is the treatment success ratio in the group of the reference drug – placebo (R, reference);

d is the superiority margin in the test and reference drug groups. d margin is 5.0%.

To test the null hypothesis a one-tailed 95% confidence interval (CI) for the ratio difference will be calculated by the method suggested in **Newcombes Hybrid Score** 

#### interval 1998.1

It is assumed that if the lower boundary of the *one-tailed* 95% CI is > d (5.0%), then the null hypothesis is rejected and an alternative hypothesis is accepted: "the test drug (Seroguard at the dose of XX) is not superior to the reference drug (placebo) by the primary endpoint".

#### 10.2 SECONDARY EFFICACY VARIABLES

## The analysis is performed only in the ITT population.

A point of "last observation" will be additionally determined for secondary efficacy variables. It is the last measurement of the parameter except the baseline (Visit 0).

The number of hyperechoic linear lesions post surgery is presented in the similar way as for the primary efficacy variable but a non-parametric Mann-Whitney test for the intergroup comparison will be calculated additionally.

Thickness of adhesions, their extent, limited mobility of pelvic organs and absence of ultrasound signs of pelvic adhesive disease will be described as nominal data. Intergroup comparisons at visits will be performed by means of the Fisher's exact test (in comparison with the placebo group). Tables will show a change in frequencies from the baseline (screening). The significance of intra-group changes will be tested by means of the symmetry test (Bowker test).

Severity of adhesions (PAI index) will be described by treatment groups and visits as a continuous value. Visit 0 (screening) is taken as the baseline. A change from the baseline also will be presented in a table. The intergroup comparison will be performed by means of a linear mixed model where a study centre is a random factor. A baseline is to be included in the model for "change in the adhesion thickness" variable (adhesion thickness at the baseline). "Seroguard, 1.5 mL/kg" and "Seroguard. 2.4 mL/kg" treatment groups will be compared to the placebo group. A Mann-Whitney test will be calculated to confirm the intergroup comparisons.

#### Adjustments for multiple comparison won't be provided.

#### 11. SAFETY ANALYSIS

# Safety analysis is performed in the safety population.

A point of "last observation" will be additionally determined for safety parameters. It is the last measurement of a parameter, including the one at the early termination visit, except the baseline (Visit 0).

#### Evaluated parameters:

- Incidence of adverse events and/or serious adverse events in the treatment groups;
- Complete blood count;
- Blood biochemistry;
- Urinalysis;
- Coagulogram;
- Concomitant therapy;
- Vital signs (body weight, blood pressure, heart rate, RR, and body temperature);
- Pregnancy test;

-

<sup>&</sup>lt;sup>11</sup> Lower boundary

- 12-lead ECG:
- Physical examination parameters;
- Abdominal ultrasound;
- Postoperative wound assessment (local status).

**Adverse event** is any untoward symptom or condition that developed after administration of a study drug even if it is not considered as having a causal relationship with this treatment. A notion of the study drug includes both the investigational product and the reference drug.

A serious adverse event is any untoward symptom or pathological condition that:

- results in death;
- 2. is life-threatening;
- 3. requires hospitalization or prolongation of existing hospitalization;
- 4. results in persistent or significant disability and/or incapacity;
- 5. results in a congenital anomaly or birth defect;
- 6. is considered to be an important medical event.

The following cases of hospitalization are not considered as serious adverse events:

- routine treatment or monitoring of the study disease if it is not related with any deterioration in the patient's condition;
- pre-planned treatment for a concurrent condition that has been diagnosed before the study initiation, is not related to the study disease, and is not worsening;
- hospitalization for general health problems not related with any deterioration in the patient's condition.

#### 11.1 ASSESSMENT OF ADVERSE EVENTS AND SERIOUS ADVERSE EVENTS

All adverse events (AEs) documented in the Case Report Forms (CRF) will be divided into TESS (events emerging during the trial, i.e. after the start of treatment) and non-TESS (see Section 6).

All adverse events will be coded by the MedDRA dictionary.

The number and percentage of patients with TESS AEs in each treatment group will be presented in tables by the system organ class and preferred term, casual relation to the study drug and degree of severity.

Treatment arms will be compared by TESS AE rates in the "system of organs" groups.

The methodology of comparison is described in:

- Helmut Strasser & Christian Weber (1999). On the asymptotic theory of permutation statistics. **Mathematical Methods of Statistics** \*8\*, 220-250.
- Torsten Hothorn, Kurt Hornik, Mark A. van de Wiel & Achim Zeileis (2006). A Lego System for Conditional Inference. **The American Statistician**, \*60\*(3), 257-263.
- Torsten Hothorn, Kurt Hornik, Mark A. van de Wiel & Achim Zeileis (2008). Implementing a class of permutation tests: The coin package, **Journal of Statistical Software**, \*28\*(8), 1-23. http://www.jstatsoft.org/v28/i08

One patient can have several MedDRA SOC (System Organ Class) terms. The number of patient's SOC terms will be counted and recorded in the matrix. If a patient has no SOC term, it is scored as "0".

# A patient's record will be presented like the following:

| Patient's<br>ID | Treatment group | SOC_2 | soc_3 | SOC_4 | SOC_5 | SOC_6 |
|---|---|---|---|---|---|---|
| XXXXXXX | XXXXXXXXXXX | xx (events) | xx (events) | xx (events) | xx (events) | xx (events) |

A test for independence of two multivariate data sets is a kind of Monte Carlo simulations. The resulting p-value allows to evaluate the difference or similarity of two groups by an aggregate parameter set (SOC terms) rather than by each parameter taken separately.

All AEs and SAEs recorded in CFRs (TESS and non-TESS) will be presented in a list.

#### 11.2 LABORATORY DATA EVALUATION

Parameters will be described as discrete variables by study visits (days). The comparison of treatment groups by laboratory test parameters is not planned.

The following information will be provided additionally:

- 1) tabulated integrated listing from the database;
- 2) tabulated integrated listing representing only laboratory test abnormalities;
- 3) separate tables of laboratory data with an analysis of parameters as quantitative variables (mean, standard deviation and median).

If repeated laboratory tests (re-tests) are performed after examination at a visit, the result of the given re-test (if not omitted) will be included in the analysis instead of the one obtained at the visit. If several repeated laboratory tests are performed the last available result will be included in the analysis.

When absolute values of the parameter are analyzed, such values like "<XX1" or ">XX" (less and more than XX) will be regarded as "XX", and "NOT FOUND" – as "0".

The treatment groups will be compared by the number of laboratory test abnormalities (separately for complete blood count, blood biochemistry, etc.) by means of the Cochran-Mantel-Haenszel test (for flags of L/N/H deviations with control by the parameter).

#### 11.3 CONCOMITANT THERAPY

Concomitant therapy will be coded and presented in groups by the ATC code. The therapy will be represented in the table by two code levels: level 3 and 5 (three and five digits of the code). The comparison of groups by this parameter is not provided.

#### 11.4 ABDOMINAL ULTRASOUND

Abnormalities found at an abdominal ultrasound examination will be presented by means of descriptive statistics (as absolute and relative frequencies) by study visits and treatment groups. Treatment groups will be compared with the use of the Fisher's exact test (with no regard of abnormalities as clinically significant / insignificant).

#### 11.5 12-LEAD ECG

Abnormalities in ECG parameters will be presented by study visits by means of descriptive statistics (as absolute and relative frequencies). Treatment groups will be

-

<sup>1</sup> XX - a numeric value

compared with the use of the Fisher's exact test (with no regard of abnormalities as clinically significant / insignificant).

ECG parameters will be also presented by means of descriptive statistics (continuous data). A change from the baseline (Visit 0) will be calculated for each parameter. Treatment groups won't be compared by values determined at the visits or by parameter changes.

#### 11.6 VITAL SIGNS ASSESSMENT

Vital signs will be presented by means of descriptive statistics. A change from the baseline will be calculated for each parameter. Treatment groups won't be compared by values determined at visits or by parameter changes.

#### 11.7 PHYSICAL EXAMINATION

Physical examination results will be presented as nominal values by means of absolute and relative frequencies in tables of changes by the study time points and treatment groups. Intergroup comparisons won't be provided.

#### 11.8 POSTOPERATIVE WOUND ASSESSMENT

Results of the postoperative wound examination will be presented as nominal values by means of absolute and relative frequencies in tables of changes by the study time points and treatment groups. Intergroup comparisons won't be provided.

#### 12. INTERIM ANALYSIS

An interim analysis is not provided.

# 13. GENERAL PROVISIONS

Visit 0 (screening) is taken as the baseline.

Unless otherwise specified all statistical tests are bilateral with 5% alpha level. Unless otherwise specified all confidence intervals (CI) are two-sided 95% ones.

Unless otherwise specified continuous data are presented by a number of observations, arithmetic mean with the standard deviation, 95 % CI, median and range. The precision is one digit to the right of the decimal point.

Unless otherwise specified nominal values are described by absolute and relative frequencies. A relative frequency is calculated on the basis of the number of patients in the population under analysis rather than the number of patients at a visit (time point).

Different time periods are calculated either on the basis of physical sense or as on the date of signing the informed consent (for age, disease duration, etc).

# 14. TABLE TEMPLATES<sup>1</sup>

Table 14.1 Patient disposition

| | Seroguard, 1.5<br>mL/kg | Seroguard, 2.4<br>mL/kg | Placebo |
|---|---|---|---|
| Number of subjects enrolled | xx (100.0%) | xx (100.0%) | xx (100.0%) |
| Safety population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| PP population | XX ( XX.X%) | xx ( xx.x%) | xx ( xx.x%) |
| ITT population | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Study completion | | | |
| Study was completed as per protocol | xx ( xx.x%) | XX ( XX.X%) | xx ( xx.x%) |
| Study was not completed | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Adverse event | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| Death | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |
| No contact with the patient | xx ( xx.x%) | xx ( xx.x%) | xx ( xx.x%) |

Table 14.2 Reasons of patients exclusion from the PP population<sup>2</sup>

| | Seroguard, 1.5<br>mL/kg | Seroguard,<br>2.4 mL/kg | Placebo |
|---|---|---|---|
| Violation of the inclusion/non-inclusion criteria | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Patient's noncompliance <sup>3</sup> | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 14.3 Reasons of patients exclusion from the ITT population Same as in Table 14.2

#### 14.1 Demographic and Other Baseline Characteristics

Table 14.4 Demographic and Other Baseline Characteristics. Screening. ITT population. N = XX

| Parameter | Seroguard,<br>1.5 mL/kg,<br>N=XX | Seroguard,<br>2.4 mL/kg,<br>N=XX | Placebo<br>N = xx | p-value |
|---|---|---|---|---|
| Age (years) | | | | 0.xxx <sup>4</sup> |
| И | XX | XX | XX | |
| Mean (SD) <sup>5</sup> | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] | |
| Median | XX.X | XX.X | XX.X | |
| Min - Max | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx | |
| Sex | | | | |
| Female | xx (100.0%) | xx (100.0%) | xx (100.0%) | |
| Race | | | | |
| Caucasian | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | |
| Other | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | |
| No data | xx (xx.x%) | xx (xx.x%) | XX (XX•X8) | |
| Height (cm) | | | | |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | XX.X (XX.X) | xx.x (xx.x) | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] | |
| Median | XX.X | XX.X | XX.X | |
| Min - Max | xx.x - xx.x | XX.X - XX.X | xx.x - xx.x | |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx | |
| Weight (kg) | | | | |
| И | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] | |
| Median | XX.X | XX.X | XX.X | |
| Min - Max | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |

<sup>&</sup>lt;sup>1</sup> Tables in the report can differ from the templates if it does not result in a loss of meaning or required information.


<sup>&</sup>lt;sup>2</sup> One patient can have several protocol violations.

<sup>&</sup>lt;sup>3</sup> If there is such a parameter

 $<sup>^{4}</sup>$  ANOVA (mixed model).  $H_{0}$ :  $\mu_{1}=\mu_{2}=\mu_{3}$ 

<sup>&</sup>lt;sup>5</sup> Standard deviation

| Parameter | Seroguard,<br>1.5 mL/kg,<br>N=XX | Seroguard,<br>2.4 mL/kg,<br>N=XX | Placebo<br>N = xx | p-value |
|---|---|---|---|---|
| p normal distribution | 0.xxx | 0.xxx | 0.xxx | |
| BMI (kg/m²) | | | | $0.xxx^1$ |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] | |
| Median | XX.X | XX.X | XX.X | |
| Min - Max | xx.x - xx.x | xx.x - xx.x | XX.X - XX.X | |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx | |

**Table 14.5** Data on disease. Screening. ITT population. N = xx

| arameter | Seroguard,<br>1.5 mL/kg | Seroguard,<br>2.4 mL/kg | Placebo<br>N = xx | p-value |
|---|---|---|---|---|
| | N = xx | N = xx | 11 - AA | 100 |
| ime since diagnosis (months) | | | | 0.xxx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] | |
| Median | XX.X | XX.X | XX.X | |
| Min - Max | XX.X - XX.X | XX.X - XX.X | XX.X - XX.X | |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx | |
| ynecological history | | | | |
| Age at menarche (years) | | | | 0.xx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] | |
| Median | XX.X | XX.X | XX.X | |
| Min - Max | xx.x - xx.x | XX.X - XX.X | XX.X - XX.X | |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx | |
| Character of menstruation | | | | 0.xx |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Abnormal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Time since last menstruation (da | ys) | | | 0.xx: |
| И | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] | |
| Median | XX.X | XX.X | XX.X | |
| Min - Max | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx | |
| Previous pregnancies | | | | 0.xx |
| No data | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Yes | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | |
| Number of pregnancies | - | | | 0.xx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] | |
| Median | XX.X | XX.X | XX.X | |
| Min - Max | XX.X - XX.X | XX.X - XX.X | xx.x - xx.x | |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx | |
| Pregnancies that resulted in bir | th (% of the total | number) | | 0.xx |
| N | XX | XX | XX | |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] | |
| Median | XX.X | XX.X | XX.X | |
| Min - Max | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x | |

 $<sup>^1</sup>$  ANOVA (mixed model).  $H_0$ :  $\mu_1=\mu_2=\mu_3$   $^2$  ANOVA (mixed model).  $H_0$ :  $\mu_1=\mu_2=\mu_3$   $^3$  ANOVA (mixed model).  $H_0$ :  $\mu_1=\mu_2=\mu_3$ 

<sup>&</sup>lt;sup>4</sup> Fisher's exact test

<sup>&</sup>lt;sup>5</sup>ANOVA (mixed model).  $H_0$ :  $\mu_1=\mu_2=\mu_3$ 

<sup>&</sup>lt;sup>6</sup> Fisher's exact test

<sup>&</sup>lt;sup>7</sup>ANOVA (mixed model).  $H_0$ :  $\mu_1=\mu_2=\mu_3$  8 ANOVA (mixed model).  $H_0$ :  $\mu_1=\mu_2=\mu_3$ 

| Parameter | Seroguard,<br>1.5 mL/kg<br>N = xx | Seroguard,<br>2.4 mL/kg<br>N = xx | Placebo<br>N = xx | p-value |
|---|---|---|---|---|
| p normal distribution | 0.xxx | 0.xxx | 0.xxx | |
| Gestation course | | | | $0.xxx^1$ |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Abnormal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Gynecological examination | 7171 (7171-710) | AM (AM•MO) | 777 (777-77-0) | |
| Mucous membrane, vagina and uterus | | | | |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Color 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Color 2 | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | |
| Type of vaginal discharge | XX (XX.XT) | XX (XX.XT) | XX (XX.X6) | |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| | 3 3 | | , , | |
| Type 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Type 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | - 0 |
| Cervix shape | , | | | 0.xxx <sup>2</sup> |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Conical | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Cylindrical | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Deformed | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| External os shape | | | | $0.xxx^3$ |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Round | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Split | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Abnormalities | | | | 0.xxx <sup>4</sup> |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| No | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Yes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Scars | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | |
| Polyps | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Ectropion | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Other | AND ALDER AND ALDERSON OF A | | AND A STATE OF A STATE | |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0 5 |
| Colposcopy | | 2 22 | | 0.xxx <sup>5</sup> |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Abnormal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Clinically insignificant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Cervical cytology by Pap smears | | | | 0.xxx <sup>6</sup> |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Abnormal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Clinically insignificant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Smear microscopy (culture test) | | | | 0.xxx <sup>7</sup> |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Normal | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | |
| Abnormal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Clinically significant | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | |
| Clinically insignificant | | | | |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Hysterosalpingography | | / | | |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Normal | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | |
| Abnormal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Clinically insignificant | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | |

<sup>&</sup>lt;sup>1</sup> Fisher's exact test

<sup>&</sup>lt;sup>2</sup> Fisher's exact test <sup>3</sup> Fisher's exact test

Fisher's exact test (yes, no, no data)
 Fisher's exact test (with no regard of data as clinically significant/insignificant)
 Fisher's exact test (with no regard of data as clinically significant/insignificant)
 Fisher's exact test (with no regard of data as clinically significant/insignificant)

Table 14.6 Previous diseases. ITT population. Screening. N = XX

| System Organ Class Term<br>Preferred Term | Seroguard, 1.5 mL/kg<br>N = xx | Seroguard, 2.4 mL/kg<br>N = xx | Placebo<br>N = xx |
|---|---|---|---|
| Patients in total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| SOC term | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 14.7 Concurrent diseases. ITT population. Screening. N = XX Same as in Table 14.6

Table 14.8 Prior therapy. Screening. ITT population. N = XX

| Therapeutic subgroup<br>Drug (ATC code) | Seroguard, 1.5<br>mL/kg<br>N = xx | Seroguard, 2.4<br>mL/kg<br>N = xx | Placebo<br>N = xx |
|---|---|---|---|
| Therapeutic subgroup (level 3 ATC code) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| Drug 1 (level 5 ATC code) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Drug 2 (level 5 ATC code) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| J.,. | | | |

Table 14.9 Physical examination. ITT population. Screening. N = xx

| Table 14.5 Fily | Sical examination. | rable 14.9 Physical examination. 111 population. Screening. N – XX | | |
|---|---|---|---|---|
| Parameter | Seroguard,<br>1.5 mL/kg<br>N = xx | Seroguard,<br>2.4 mL/kg<br>N = xx | Placebo<br>N = xx | p-value |
| General health | | | | $0.xxx^1$ |
| Not assessed/ no data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Abnormal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Clinically significant | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Clinically insignificant | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | |
| No data | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | |
| Skin | | | | |
| Musculoskeletal system | | | | |
| Lymph nodes | | | | |
| Thyroid | | | | |
| Upper airways | | | | |
| Lungs | | | | |
| Cardiovascular system | | | | |
| Abdominal organs | | | | |
| Kidneys | | | | |
| Mental status | | | | |
| - 1000 | | | The state of the s | |


<sup>&</sup>lt;sup>1</sup> Cochran-Mantel-Haenszel test (for flags of Normal/Abnormal/No data with control by the parameter)

**Table 14.10** HIV, RW, HBV and HCV test results. ITT population. N = XX

| Parameter | Seroguard, 1.5 mL/kg<br>N = xx | Seroguard, 2.4 mL/kg<br>N = xx | Placebo<br>N = xx |
|---|---|---|---|
| HIV | | | |
| (-) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| (+) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| RW | | | |
| (-) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| (+) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| HBV | | | |
| (-) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| (+) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| HCV | | | |
| (-) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| (+) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

**Table 14.11** Pregnancy test. Screening. ITT population. N = XX

| Parameter | Seroguard,<br>1.5 mL/kg<br>N = xx | Seroguard,<br>2.4 mL/kg<br>N = xx | Placebo<br>N = xx |
|---|---|---|---|
| Pregnancy test | | i e | |
| Negative | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Positive | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| No data/not performed | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |

**Table 14.12** 12-lead ECG Screening. ITT population. N = XX

| Group | Normal | Abnor Clinically | | No data | p-value <sup>1</sup> |
|---|---|---|---|---|---|
| 12-lead ECG | | | | | 0.xxx |
| Seroguard, 1.5 mL/kg | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Seroguard, 2.4 mL/kg | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | |
| Placebo | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

**Table 14.13** Vital signs. ITT population. Screening. N = XX

| | Result | | | | |
|---|---|---|---|---|---|
| Group | Normal | Abnor Clinically insignificant | Clinically | No data | p-value <sup>2</sup> |
| RR | 1 | Indignitionne | DIGHTLICANC | | 0.xxx |
| Seroguard, 1.5 mL/kg | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Seroguard, 2.4 mL/kg | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Placebo | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| HR | | | | | |
| 1 | | | | | |

Parameters: RR, HR, SBP, DBP, body temperature.


<sup>&</sup>lt;sup>1</sup> Fisher's exact test (with no regard of data as clinically significant/insignificant) <sup>2</sup> Fisher's exact test (with no regard of data as clinically significant/insignificant)

# 14.2 EFFICACY ANALYSIS

# 14.2.1 Primary efficacy variable

Table 14.14 Treatment success. Decrease in the number of adhesions. ITT population. N = XX

| Parameter | Seroguard,<br>1.5 mL/kg<br>N = xx | Seroguard,<br>2.4 mL/kg<br>N = xx | Placebo<br>N = xx |
|---|---|---|---|
| Treatment success (reduction of the adhesions number by 3 or more) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| $p_T - p_R$ 95% CI [xx.x;] | x.xx [xx.x;] | x.xx [xx.x;] | |

Table 14.15 Treatment success. Decrease in the number of adhesions. PP population. N = XX

| Parameter | Seroguard,<br>1.5 mL/kg<br>N = xx | Seroguard,<br>2.4 mL/kg<br>N = xx | Placebo<br>N = xx |
|---|---|---|---|
| Treatment success (reduction of the adhesions number by 3 or more) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| $p_T - p_R$ 95% CI [xx.x;] | x.xx [xx.x;] | x.xx [xx.x;] | |

# 14.2.2 Secondary efficacy variables

Table 14.16 Assessment of adhesion severity by PAI (Pelvic Adhesions Index) ITT population. N = XX

| | Seroguard, | Seroguard, | Placebo |
|---|---|---|---|
| Parameter | 1.5 mL/kg | 2.4 mL/kg | N = xx |
| | N = xx | N = xx | 14 - XX |
| Visit 0 (Screening). Baseline | | | |
| И | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] |
| Median | XX.X | XX.X | XX.X |
| Min - Max | xx.x - xx.x | xx.x - xx.x | XX.X - XX.X |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx |
| p-ANOVA vs.¹ Placebo | 0.xxx/0.xxx | 0.xxx/0.xxx | |
| Visit 3 (day 30±4). Observation | | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] |
| Median | XX.X | XX.X | XX.X |
| Min - Max | XX.X - XX.X | XX.X - XX.X | XX.X - XX.X |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx |
| p-ANOVA vs.² Placebo | 0.xxx/0.xxx | 0.xxx/0.xxx | |
| Change. Visit 3 (day 30±4). Observ | ation | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] |
| Median | XX.X | XX.X | XX.X |
| Min - Max | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx |
| p-value for change | 0.xxx | 0.xxx | 0.xxx |
| p-ANOVA vs.³ Placebo | 0.xxx/0.xxx | 0.xxx/0.xxx | |
| Early termination visit (last avai | lable observation) | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] |
| Median | XX.X | XX•X | XX.X |
| Min – Max | XX•X - XX•X | XX•X - XX•X | XX.X - XX.X |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx |
| p-ANOVA vs.4 Placebo | 0.xxx/0.xxx | 0.xxx/0.xxx | |
| p-ANOVA vs.4 Placebo<br>Change. Early termination visit (1 | | | ζ. |

<sup>&</sup>lt;sup>1</sup> ANOVA (mixed model) / Mann-Whitney test


<sup>&</sup>lt;sup>2</sup> ANOVA (mixed model) / Mann-Whitney test

<sup>&</sup>lt;sup>3</sup> ANOVA (mixed model) / Mann-Whitney test

<sup>&</sup>lt;sup>4</sup> ANOVA (mixed model) / Mann-Whitney test

| Parameter | Seroguard,<br>1.5 mL/kg<br>N = xx | | Placebo<br>N = xx |
|---|---|---|---|
| N | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] |
| Median | XX.X | XX.X | XX.X |
| Min - Max | XX.X - XX.X | XX.X - XX.X | XX.X - XX.X |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx |
| p-value for change | 0.xxx | 0.xxx | 0.xxx |
| p-ANOVA vs.¹ Placebo | 0.xxx/0.xxx | 0.xxx/0.xxx | |

Number of hyperechoic linear lesions post surgery as based on transvaginal ultrasound results. ITT population. N = XX**Table 14.17** 

| | · · | | |
|---|---|---|---|
| Parameter | Seroguard,<br>1.5 mL/kg | Seroguard,<br>2.4 mL/kg | Placebo<br>N = xx |
| | N = xx | N = xx | N - XX |
| Visit 0 (Screening) Baseline | | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] |
| Median | XX.X | XX.X | XX.X |
| Min - Max | XX.X - XX.X | xx.x - xx.x | $XX \cdot X - XX \cdot X$ |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx |
| p-ANOVA vs.2 Placebo | 0.xxx/0.xxx | 0.xxx/0.xxx | |
| Visit 3 (day 30±4). Observation | | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] |
| Median | XX.X | XX•X | XX.X |
| Min - Max | xx.x - xx.x | xx.x - xx.x | XX.X - XX.X |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx |
| p-ANOVA vs.³ Placebo | 0.xxx/0.xxx | 0.xxx/0.xxx | |
| Change. Visit 3 (day 30±4). Obse | rvation | - | |
| N | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] |
| Median | XX.X | XX.X | XX.X |
| Min - Max | xx.x - xx.x | xx.x - xx.x | xx.x - xx.x |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx |
| p-value for change | 0.xxx | 0.xxx | 0.xxx |
| p-ANOVA vs.4 Placebo | 0.xxx/0.xxx | 0.xxx/0.xxx | |
| Early termination visit (last av | ailable observation) | | |
| N | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] |
| Median | XX.X | XX.X | XX.X |
| Min - Max | xx•x - xx•x | xx.x - xx.x | xx.x - xx.x |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx |
| p-ANOVA vs.5 Placebo | 0.xxx/0.xxx | 0.xxx/0.xxx | |
| Change. Early termination visit | (last available observation | on) | |
| N | XX | XX | XX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| 95% CI | [xx.x; xx.x] | [xx.x; xx.x] | [xx.x; xx.x] |
| Median | XX.X | XX.X | XX.X |
| Min - Max | xx.x - xx.x | xx.x - xx.x | XX.X - XX.X |
| p normal distribution | 0.xxx | 0.xxx | 0.xxx |
| p-value for change | 0.xxx | 0.xxx | 0.xxx |
| p-ANOVA vs.6 Placebo | 0.xxx/0.xxx | 0.xxx/0.xxx | |

<sup>&</sup>lt;sup>1</sup> ANOVA (mixed model) / Mann-Whitney test <sup>2</sup> ANOVA (mixed model) / Mann-Whitney test <sup>3</sup> ANOVA (mixed model) / Mann-Whitney test <sup>4</sup> ANOVA (mixed model) / Mann-Whitney test <sup>5</sup> ANOVA (mixed model) / Mann-Whitney test <sup>6</sup> ANOVA (mixed model) / Mann-Whitney test

Table 14.18 Limited mobility of pelvic organs post surgery. ITT population. N = XX

| Parameter | Seroguard,<br>1.5 mL/kg<br>N = xx | Seroguard, $2.4 \text{ mL/kg}$ $N = xx$ | Placebo<br>N = xx |
|---|---|---|---|
| Visit 0 (Screening) | | | |
| Detected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not detected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No data <sup>1</sup> | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value (Fisher's test) vs. Placebo | 0.xxx | 0.xxx | |
| Visit 3 (day 30±4). Observation | | | |
| Detected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not detected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value (Fisher's test) vs. Placebo | 0.xxx | 0.xxx | |
| Early termination visit (last available observation) | | | |
| Detected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not detected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value (Fisher's test) vs. Placebo | 0.xxx | 0.xxx | |

| Visit 0 (Screening) | Se: | Visit 3 (day 30±4). Observation Seroguard, 1.5 mL/kg Seroguard, 2.4 mL/kg Placebo N = xx N = xx | | | | d, 1.5 mL/kg Seroguard, 2.4 mL/kg Placebo | | | Total | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Detected | Not detected | No data | Detected | Not detected | No data | Detected | Not detected | No data | |
| Detected | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) |
| Not detected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No data <sup>2</sup> | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-Bowker's | | 0.xxx | | | 0.xxx | | | 0.xxx | | |

| | Early termination visit (last available observation) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit 0 (Screening) | Seroguard, 1.5 mL/kg N = xx | | Seroguard, 2.4 mL/kg $N = xx$ | | Placebo<br>N = xx | | | Total | | |
| | Detected | Not detected | No data | Detected | Not detected | No data | Detected | Not detected | No data | |
| Detected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not detected | xx (xx,x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| No data <sup>3</sup> | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-Bowker's | | 0.xxx | | | 0.xxx | | | 0.xxx | | |

<sup>&</sup>lt;sup>1</sup> If the data set is complete this category should be omitted

<sup>&</sup>lt;sup>2</sup> If the data set is complete this category should be omitted <sup>3</sup> If the data set is complete this category should be omitted

Table 14.19 Absence of pelvic adhesive disease signs. ITT population. N = XX

| Parameter | Seroguard, 1.5 mL/kg $N=xx$ | Seroguard, 2.4 mL/kg<br>N = xx | Placebo<br>N = xx |
|---|---|---|---|
| Visit 0 (Screening) | | | |
| None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Detected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No data¹ | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value (Fisher's test) vs. Placebo | 0.xxx | 0.xxx | |
| Visit 3 (day 30±4). Observation | | | |
| None | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| Detected | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value (Fisher's test) vs. Placebo | 0.xxx | 0.xxx | |
| Early termination visit (last available observation) | | | |
| None | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| Detected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value (Fisher's test) vs. Placebo | 0.xxx | 0.xxx | |

| Visit 0 (Screening) | Ser | oguard, 1.5 mL/<br>N = xx | ′kg | | (day 30±4). Obs<br>coguard, 2.4 mL/<br>N = xx | | | Placebo<br>N = xx | | Total |
|---|---|---|---|---|---|---|---|---|---|---|
| | None | Detected | No data | None | Detected | No data | None | Detected | No data | |
| None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Detected | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) |
| No data <sup>2</sup> | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) |
| Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-Bowker's | | 0.xxx | | | 0.xxx | | | 0.xxx | | |

| | | | Early t | ermination vi | sit (last ava | ilable obser | vation) | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Visit 0 (Screening) | Ser | oguard, 1.5 mL/ $N = xx$ | 'kg | Ser | roguard, 2.4 $mL$ / $N = xx$ | 'kg | | Placebo<br>N = xx | | Total |
| | None | Detected | No data | None | Detected | No data | None | Detected | No data | |
| None | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) |
| Detected | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| No data³ | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-Bowker's | | 0.xxx | | | 0.xxx | | | 0.xxx | | |

<sup>&</sup>lt;sup>1</sup> If the data set is complete this category should be omitted

<sup>&</sup>lt;sup>2</sup> If the data set is complete this category should be omitted <sup>3</sup> If the data set is complete this category should be omitted

Table 14.20 Thickness of adhesions. ITT population. N = XX

| Parameter | Seroguard, 1.5 mL/kg $N = xx$ | Seroguard, 2.4 mL/kg<br>N = xx | Placebo<br>N = xx |
|---|---|---|---|
| Visit 0 (Screening) | | | |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 0* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1* | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| 2* | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| 3* | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| p-value (Fisher's test) vs. Placebo | 0.xxx | 0.xxx | |
| Visit 3 (day 30±4). Observation | | | |
| No data | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| 0* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value (Fisher's test) vs. Placebo | 0.xxx | 0.xxx | |
| Early termination visit (last available observation) | | | |
| No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 0* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 3* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| p-value (Fisher's test) vs. Placebo | 0.xxx | 0.xxx | |

\*0 - none; 1 - thin; 2 - marked; 3- marked with an impaired passage through organs involved.

| | | | | Visit 3 (day 30 | )±4) | | |
|---|---|---|---|---|---|---|---|
| roup | Visit 0 (Screening) | No data | 0* | 1* | 2* | 3* | Total |
| | No data | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 0* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 1* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| _ | 2* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| λg | 3* | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| મું | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | жж (жж.ж <del>8</del> ) |
| ь<br>Г | p-value1 | 0.xxx | | | | | |
| -: | | | | | | | |
| <del>-</del> | | | | | | | |
| | | | | Last observatio | n/study completion d | ate | |
| | Visit 0 (Screening) | No data | 0* | Last observatio | on/study completion d | ate<br>3* | Total |
| | Visit 0 (Screening) No data | <b>No data</b> xx (xx.x%) | 0*<br>xx (xx.x%) | | | AND THE PARTY OF T | Total<br>xx (xx.x%) |
| | | | | 1* | 2* | 3* | |
| eroguard, 1. | No data | xx (xx.x%) | xx (xx.x%) | 1*<br>xx (xx.x%) | 2*<br>xx (xx.x%) | 3*<br>xx (xx.x%) | xx (xx.x%) |
| | No data<br>0* | xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) | 1*<br>xx (xx.x%)<br>xx (xx.x%) | 2* xx (xx.x%) xx (xx.x%) | 3*<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%) |
| eroguard, 1. | No data<br>0*<br>1* | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | 1* | 2* | 3* xx (xx.x%) xx (xx.x%) xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) |
| eroguard, 1. | No data<br>0*<br>1*<br>2* | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%)<br>xx (xx.x%) | 1* | 2* | 3* | xx (xx.x8)<br>xx (xx.x8)<br>xx (xx.x8) |

<sup>1</sup> p-Bowker

| SG-2/1215 Statisti | ical Analysis Plan | | Final version 1.2 | | | | |
|---|---|---|---|---|---|---|---|
| Group | Visit 0 (Screening) | No data | 0* | Visit 3 (day 30±4)<br> 1* | 2* | 3* | Total |
| Seroguard, 2.4<br>mL/kg | | | | | | | |

Table 14.21 Extent of the adhesion process in the pelvic cavity. ITT population. N = XX Same as in Table 14.20

\*0 - none; 1 - one region (right lateral space, left lateral space, Douglas pouch or vesicouterine pouch); 2 - two regions; 3 - subtotal pelvic adhesions (three regions); 4 - total pelvic adhesions.

#### 14.3 SAFETY ANALYSIS

Placebo

Table 14.22 12-lead ECG during the study. Safety population. N = XX

| | | | Res<br>Abno | | | |
|---|---|---|---|---|---|---|
| Group | Visit | Normal | Clinically<br>insignificant | Clinically<br>significant | No data | p-value |
| 12-lead ECG | | | | | | |
| Seroguard, 1.5 mL/kg | Visit 0 (Screening) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | 0.xxx |
| Seroguard, 2.4 mL/kg | Visit 0 (Screening) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | |
| Placebo | Visit 0 (Screening) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | |
| Seroguard, 1.5 mL/kg | Visit 2 (day 6±1) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Seroguard, 2.4 mL/kg | Visit 2 (day 6±1) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Placebo | Visit 2 (day 6±1) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | |
| Seroguard, 1.5 mL/kg | Visit 3 (day 30±4) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | 0.xxx |
| Seroguard, 2.4 mL/kg | Visit 3 (day 30±4) | XX (XX.X%) | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | |
| Placebo | Visit 3 (day 30±4) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | |
| Seroguard, 1.5 mL/kg | Last observation/study completion<br>date | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Seroguard, 2.4 mL/kg | Last observation/study completion<br>date | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Placebo | Last observation/study completion date | xx (xx.x%) | xx (xx.x%) | xx (xx.x8) | xx (xx.x%) | |

<sup>&</sup>lt;sup>1</sup> p-Bowker

<sup>&</sup>lt;sup>2</sup> Fisher's exact test (with no regard of data as clinically significant/insignificant)

Table 14.23 12-lead ECG during the study. Absolute values. Safety population. N = XX

| | Froup Visit | | | Result | | | | | | | C | hange | | | p-value | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | Visit | | Mean | SD | Median | Min. | Max. | Norm. | | Mean | SD | Median | Min. | Max. | Norm. | Change |
| HR (beats per minute) | <u> </u> | | | | | | | | | - 1 | * | - | | <i>-</i> | ė. | |
| Seroguard, 1.5mL/kg | Visit 0 (Screening) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | | | | | | | | |
| Seroguard, 2.4mL/kg | Visit O (Screening) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | | | | | | | | |
| Placebo | Visit O (Screening) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | | | | | | | | |
| Seroguard, 1.5mL/kg | Visit 2 (day 6±1) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| Seroguard, 2.4mL/kg | Visit 2 (day 6±1) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| Placebo | Visit 2 (day 6±1) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| PR (ms) | · | | | | | | | | | | | | | | | |

Parameters: HR, PR, QRS, QT, QTc

Table 14.24 Abdominal ultrasound during the study. Safety population. N = XX

| Froup | Visit | Normal | Clinically<br>insignificant | | No data | p-value <sup>1</sup> |
|---|---|---|---|---|---|---|
| Abdominal ultrasound | | | | | | |
| Seroguard, 1.5 mL/kg | Visit 0 (Screening) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Seroguard, 2.4 mL/kg | Visit 0 (Screening) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | |
| Placebo | Visit 0 (Screening) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | XX (XX.X%) | |
| Seroguard, 1.5 mL/kg | Visit 2 (day 6±1) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | XX (XX.X%) | 0.xxx |
| Seroguard, 2.4 mL/kg | Visit 2 (day 6±1) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Placebo | Visit 2 (day 6±1) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Seroguard, 1.5 mL/kg | Last observation/study<br>completion date | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Seroguard, 2.4 mL/kg | Last observation/study<br>completion date | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |
| Placebo | Last observation/study completion date | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | |

<sup>&</sup>lt;sup>1</sup> Fisher's exact test (with no regard of data as clinically significant/insignificant)

Table 14.25 Physical examination. Safety population. N = xx

| | | | | | Result | | |
|---|---|---|---|---|---|---|---|
| | | | | Abnormal finding | Result | | |
| Group | Visit | Parameter | No data | Clinically insignificant | Clinically<br>significant | Normal | Not assessed/ no<br>data |
| _ | ' | General health | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| mL/kg | | Skin | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ę | | Musculoskeletal system | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 5 | | Lymph nodes | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| i i | | Thyroid | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Upper airways | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, | | Lungs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Z<br>a | | Cardiovascular system | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| <b>6</b> 0 | | Abdominal organs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 9 | | Kidneys | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 02 | | Mental status | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 770 | 0 | General health | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| mL/kg | Бау | Skin | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ē, | Õ | Musculoskeletal system | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 4 I | Z | Lymph nodes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | Surgery | Thyroid | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1.7 | ŭ | Upper airways | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| eroguard, | Ø | Lungs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Па | ÷ | Cardiovascular system | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 0, | 4 | Abdominal organs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Ser | ω<br>- Η | Kidneys | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 01 | _ :5 | Mental status | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | General health | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Skin | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Musculoskeletal system | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 0 | | Lymph nodes | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| pde | | Thyroid | XX (XX.X8) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ů<br>G | | Upper airways | XX (XX.X%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Placebo | | Lungs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Cardiovascular system | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Abdominal organs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Kidneys | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Mental status | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 14.26 Local status assessment. Safety population. N = XX

| | | | | Result | |
|---|---|---|---|---|---|
| Group | Visi | Parameter | No data | No | Yes |
| Seroguard, 1.5 mL/kg | | Tenderness on palpation | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| | | Hyperemia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 1 | Oedema | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | <del>+</del> 9 | Exudate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 2.4 mL/kg | Σ | Tenderness on palpation | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| | (day | Hyperemia | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| | 01 | Oedema | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | 11 | Exudate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Placebo | 110 | Tenderness on palpation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Ϋ́, | Hyperemia | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Oedema | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | Exudate | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 14.27 Pregnancy test. Safety population. N = XX

| | | | Result | |
|---|---|---|---|---|
| Group | Visit | Negative | Positive | Not<br>assessed/<br>no data |
| Seroguard, 1.5 mL/kg | Visit 0. Screening | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 2.4 mL/kg | Visit O. Screening | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Placebo | Visit O. Screening | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 1.5<br>mL/kg | Visit 3. Day 30±4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 2.4<br>mL/kg | Visit 3. Day 30±4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Placebo | Visit 3. Day 30±4 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 1.5<br>mL/kg | Last observation/ Study completion | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 2.4<br>mL/kg | Last observation/ Study completion | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) |
| Placebo | Last observation/ Study completion | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

Table 14.28 Concomitant therapy during the study. Safety population. N = XX

| Therapeutic subgroup<br>Drug (ATC code) | Seroguard,<br>1.5 mL/kg<br>N = xx | Seroguard,<br>2.4 mL/kg<br>N = xx | Placebo<br>N = xx |
|---|---|---|---|
| Therapeutic subgroup (level 3 ATC code) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Drug 1 (level 5 ATC code) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) |
| Drug 2 (level 5 ATC code) | xx (xx.x%) | XX (XX.X%) | XX (XX.X%) |

Table 14.29 Vital signs. Safety population. N = XX

| | | | | | | 2007 | 1007 | 1017 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Group Visit | | | | | Result | | | | | | C | hange | | | <i>y</i> −q | value |
| GLOUP | VISIC | | Mean | SD | Median | Min. | Max. | Norm. | | Mean | SD | Median | Min. | Max. | Norm. | Change |
| HR (beats per minute) | | 111 | 100 | <u> </u> | | | 4 | · · | | | <i>'</i> | | - 12 | No. | | |
| Seroguard, 1.5 mL/kg | Visit 0 (Screening) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | | | | | | | | |
| Seroguard, 2.4 mL/kg | Visit 0 (Screening) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | | | | | | | | |
| Placebo | Visit 0 (Screening) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | | | | | | | | |
| Seroguard, 1.5 mL/kg | Visit 1 (day 0) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| Seroguard, 2.4 mL/kg | Visit 1 (day 0) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| Placebo | Visit 1 (day 0) | XX. | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| RR (per minute) | | | | | | | | | | | | | | | | |

Parameters: RR, HR, SBP, DBP, body temperature.

Table 14.30 Laboratory data evaluation. Coagulogram. Safety population. N = XX

| | 14510 14.00 | East atory data | evaluation. oougule | grain Daicty | population it AA | | |
|---|---|---|---|---|---|---|---|
| | | | | Re | sult | | |
| Group | Visit | Lower tha | | | Higher than | | No data |
| | ,1520 | Clinically<br>insignificant | Clinically<br>significant | Normal | Clinically<br>insignificant | Clinically<br>significant | |
| Clotting time | | | | | | | • |
| Seroguard, 1.5 mL/kg | Visit 0 (Screening) | XX (XX.X%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 2.4 mL/kg | Visit 0 (Screening) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Placebo | Visit 0 (Screening) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 1.5 mL/kg | Visit 3 (day 30±4) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 2.4 mL/kg | Visit 3 (day 30±4) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Placebo | Visit 3 (day 30±4) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 1.5 mL/kg | Last observation/study<br>completion date | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 2.4 mL/kg | Last observation/study completion date | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Placebo | Last observation/study completion date | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Thrombin time | | | | | | | |
| INR | | | | | | | |
| APTT | | | | | | | |

Table 14.31 Laboratory data evaluation. Coagulogram. Abnormal findings only. Safety population. N = XX

| | The state of the s | | | | |
|---|---|---|---|---|---|
| | | Result | | | |
| Group | 772 - 2 4 | Lower than | normal | Higher than | n normal |
| | Visit | Clinically insignificant | Clinically<br>significant | Clinically insignificant | Clinically<br>significant |
| Clotting time | | | - | | |
| Seroguard, 1.5 mL/kg | Visit 0 (Screening) | xx (xx.x8) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 2.4 mL/kg | Visit 0 (Screening) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Placebo | Visit 0 (Screening) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

| Group | | | Result | | |
|---|---|---|---|---|---|
| | Visit | Lower tha | n normal | Higher that | an normal |
| | VISIC | Clinically | Clinically | Clinically | Clinically |
| | | insignificant | significant | insignificant | significant |
| Thrombin time | | | | | |
| INR | | | | | |
| APTT | | | | | |

Table 14.32 Laboratory data evaluation. Complete blood count. Safety population. N = XX

| | | | | Result | | | |
|---|---|---|---|---|---|---|---|
| | | Lower than | normal | | Higher tha | n normal | No data |
| Group | Visit | Clinically | Clinically | Normal | Clinically | Clinically | (36), W SALORONO. |
| | | insignificant | significant | | insignificant | significant | |
| Haemoglobin | | | | | | | •/- |
| Seroguard, 1.5 mL/kg | Visit O (Screening) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Seroguard, 2.4 mL/kg | Visit 0 (Screening) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Placebo | Visit 0 (Screening) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Seroguard, 1.5 mL/kg | Visit 2 (day 6±1) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Seroguard, 2.4 mL/kg | Visit 2 (day 6±1) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x% |
| Placebo | Visit 2 (day 6±1) | xx (xx.x%) | xx (xx.x%) | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Seroguard, 1.5 mL/kg | Visit 3 (day 30±4) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Seroguard, 2.4 mL/kg | Visit 3 (day 30±4) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Placebo | Visit 3 (day 30±4) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Seroguard, 1.5 mL/kg | Last observation/study<br>completion date | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Seroguard, 2.4 mL/kg | Last observation/study completion date | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Placebo | Last observation/study<br>completion date | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x% |
| Hematocrit | | | | | | | |
| RBC | | | | | | | |
| WBC | | | | | | | |
| Platelet count | | | | | | | |

p-value =  $0.xxx^1$ 

<sup>&</sup>lt;sup>1</sup> Cochran-Mantel-Haenszel test (for flags of L/N/H deviations with control by the parameter)

Table 14.33 Laboratory data evaluation. Complete blood count. Abnormal findings only. Safety population. N = XX

| | | | Result | | |
|---|---|---|---|---|---|
| Chair | Visit | Lower than | normal | Higher than | n normal |
| Group | Visit | Clinically | Clinically | Clinically | Clinically |
| | | insignificant | significant | insignificant | significant |
| Haemoglobin | | | | | |
| Seroguard, 1.5 mL/kg | Visit 0 (Screening) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 2.4 mL/kg | Visit 0 (Screening) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Placebo | Visit 0 (Screening) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 1.5 mL/kg | Visit 2 (day 6±1) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Seroguard, 2.4 mL/kg | Visit 2 (day 6±1) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Placebo | Visit 2 (day 6±1) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Hematocrit | | | | | |
| RBC | | | | | |
| WBC | | | | | |
| Platelet count | | | | | |

Table 14.34 Laboratory data evaluation. Blood biochemistry. Safety population. N = XX Same as in Tables 14.30, 14.32

Table 14.35 Laboratory data evaluation. Blood biochemistry. Abnormal findings only. Safety population. N = XX Same as in Tables 14.31,14.33

Table 14.36 Laboratory data evaluation. Urinalysis. Safety population. N = XX Same as in Tables 14.30, 14.32

Table 14.37 Laboratory data evaluation. Urinalysis. Abnormal findings only. Safety population. N = XX Same as in Tables 14.31,14.33

Table 14.38 Brief summary of adverse events. Safety population. N = XX

| Parameter | Seroguard,<br>1.5 mL/kg<br>N = xx | Seroguard,<br>2.4 mL/kg<br>N = xx | Placebo<br>N = XX | p-value <sup>1</sup> |
|---|---|---|---|---|
| Patients with AEs <sup>2</sup> | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Patients with SAEs <sup>3</sup> | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Patients with AE with fatal outcome | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Patients with mild to moderate AEs | XX (XX.X%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Patients with severe AEs | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Patients with AEs related or possibly related to the study drug (certain, probable, possible, unlikely, conditional or unclassifiable relation) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |
| Patients with AEs that resulted in drug withdrawal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | 0.xxx |

Table 14.39 Adverse Events. Safety population. N = XX

| MEDDRA System Organ Class term MEDDRA Preferred term | Seroguard, 1.5 m | L/kg | Seroguard, 2.4 m | L/kg | Placebo<br>n (%) | |
|---|---|---|---|---|---|---|
| rabban fletefled telm | X (%) | Y | X (%) | Y | X (%) | Y |
| Patients with AEs | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| SOC term | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred term 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred term 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |

X = number of patients who experienced at least one event of the given group.

3 SAEs only

<sup>% =</sup> percentage of patients who experienced at least one event of the given group.

Y = total number of events p-value = 0.xxx

<sup>&</sup>lt;sup>1</sup> Fisher's exact test <sup>2</sup> AEs and SAEs

Table 14.40 Serious adverse events. Safety population. N = XX

| MEDDRA System Organ Class term<br>MEDDRA Preferred term | Seroguard, 1.5 m | L/kg | Seroguard, 2.4 m | L/kg | Placebo<br>n (%) | |
|---|---|---|---|---|---|---|
| PHODINI FICIEITEG CEIM | X (%) | Y | X (%) | Y | X (%) | Y |
| Patients with SAEs | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| SOC term | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred term 1 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred term 2 | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |

X = number of patients who experienced at least one event of the given group.

Y = total number of events

Table 14.41 Adverse events by the degree of severity. Safety population. N = XX

| MEDDRA System Organ Class term MEDDRA Preferred term | Degree of | Seroguard, 1.5 mL/kg<br>n (%) | | Seroguard, 2.4 m<br>n (%) | nL/kg | Placebo<br>n (%) | |
|---|---|---|---|---|---|---|---|
| MLDDKA Freierred term | severity | X (%) | Y | X (%) | Y | X (%) | Y |
| Patients with AEs | | | | | | | |
| | Mild | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Moderate | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Severe | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| SOC term | | | | | | | |
| Preferred term 1 | Mild | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred term 2 | Mild | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Moderate | | | | | | |

X = number of patients who experienced at least one event of the given group.

Y = total number of events

 $<sup>% = % \</sup>left( {{{\mathbf{F}}_{i}}} \right)$  percentage of patients who experienced at least one event of the given group.

<sup>% =</sup> percentage of patients who experienced at least one event of the given group.

Table 14.42 Serious adverse events by the degree of severity. Safety population. N = XX

| MEDDRA System Organ Class term MEDDRA Preferred term | Degree of | Seroguard, 1.5 mL/kg n (%) | | Seroguard, 2.4 1<br>n (%) | nL/kg | Placebo<br>n (%) | |
|---|---|---|---|---|---|---|---|
| MEDDRA Freierred term | severity | X (%) | Y | X (%) | Y | X (%) | Y |
| Patients with SAEs | | | | | | | |
| | Mild | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Moderate | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Severe | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| SOC term | | | | | | | |
| Preferred term 1 | Mild | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred term 2 | Mild | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| | Moderate | | | | | | |

X = number of patients who experienced at least one event of the given group.

% = percentage of patients who experienced at least one event of the given group. Y = total number of events

Table 14.43 Adverse events and their relation to the study drug. Safety population. N = XX

| MEDDRA System Organ Class term<br>MEDDRA Preferred term | Relation to the study drug (as assessed by the investigator) | Seroguard<br>1.5 mL/kg<br>n (%) | | Seroguard<br>2.4 mL/kg<br>n (%) | | Placebo<br>n (%) | |
|---|---|---|---|---|---|---|---|
| | | X (%) | Y | X (%) | Y | X (%) | Y |
| Patients with AEs | | | | | | | |
| | Not related | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Certain | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Probable | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Possible | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Unlikely | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Conditional | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Unclassifiable | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| SOC term | | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| Preferred term 1 | Certain | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred term 2 | Unlikely | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |

X = number of patients who experienced at least one event of the given group.

% = percentage of patients who experienced at least one event of the given group.

Y = total number of events

Table 14.44 Serious adverse events and their relation to the study drug. Safety population. N = XX

| MEDDRA System Organ Class term<br>MEDDRA Preferred term | Relation to the study drug (as assessed by the investigator) | Seroguard<br>1.5 mL/kg<br>n (%) | | Seroguard<br>2.4 mL/kg<br>n (%) | | Placebo<br>n (%) | |
|---|---|---|---|---|---|---|---|
| | | X (%) | Y | X (%) | Y | X (%) | Y |
| Patients with SAEs | | | | | | | |
| | Not related | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Certain | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Probable | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Possible | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Unlikely | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Conditional | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| | Unclassifiable | xx (xx.x) | | xx (xx.x) | | xx (xx.x) | |
| SOC term | | xx (xx.x) | xx | xx (xx.x) | xx | xx (xx.x) | xx |
| Preferred term 1 | Certain | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |
| Preferred term 2 | Unlikely | xx (xx.x) | XX | xx (xx.x) | XX | xx (xx.x) | XX |

X = number of patients who experienced at least one event of the given group. % = percentage of patients who experienced at least one AE of the given group. Y = total number of events

Table 14.45 Laboratory data evaluation. Complete blood count. Absolute values. Safety population. N = XX

| Group | Visit | | | | Result | | | | | | Change | | | 0.1 | p-va | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| GLOUP | VISIT | | Mean | SD | Median | Min. | Max. | Norm. | | Mean | SD | Median | Min. | Max. | Norm. | Change |
| Haemoglobin (g/dL) | | | | | | | | | | | | | | | | |
| Seroguard, 1.5 mL/kg | Visit 0 (Screening) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | | | | | | | | |
| Seroguard, 2.4 mL/kg | Visit 0 (Screening) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | | | | | | | | |
| Placebo | Visit 0 (Screening) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | | | | | | | | |
| Seroguard, 1.5 mL/kg | Visit 2 (day 6±1) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| Seroguard, 2.4 mL/kg | Visit 2 (day 6±1) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| Placebo | Visit 2 (day 6±1) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| Seroguard, 1.5 mL/kg | Visit 3 (day 30±4) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| Seroguard, 2.4 mL/kg | Visit 3 (day 30±4) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| Placebo | Visit 3 (day 30±4) | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| Seroguard, 1.5 mL/kg | Last observation<br>/study completion<br>date | XX | XX.X | XX.X | XX,X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0,xxx |
| Seroguard, 2.4 mL/kg | Last observation<br>/study completion<br>date | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| Placebo | Last observation<br>/study completion<br>date | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | XX | XX.X | XX.X | XX.X | XX.X | XX.X | 0.xxx | 0.xxx |
| Hematocrit (%) | | | | | | | | | | | | | | | | |

# Table 14.46 Laboratory data evaluation. Blood biochemistry. Absolute values. Safety population. N = XX Same as in Table 14.45

Table 14.47 Laboratory data evaluation. Urinalysis.
Absolute values. Safety population. N = XX

Same as in Table 14.45

Table 14.48 Laboratory data evaluation. Coagulogram.
Absolute values. Safety population. N = XX

Same as in Table 14.45

Listing. 1 Adverse Events. Listing AEDDRA System Organ Class AE resolution date Degree of severity Was treatment for the AE assigned? Is the AE serious? AE starting date Low Level Term Relation to the study drug Preferred Term Centre-Patient AE description AE outcome Age (years) AE number ፷ XXXXXXX xxxxxxxxxx xxxxxxxxxxx xxxxxxxxxx XXXX XXXX xxx xxxxxx xxxx XXXXXXXXXXX XXXX XX-XXX xx-xx-xxx xx-xx-xxx XXXXXX XXXXXXX XXXXXXXXXX XXXXXXXXXX xxxxxxxxxx xxxxxxxxxx XXXX XXXX XXXX XXX xxxxxx XXXX XX-XXX xx-xx-xxx xx-xx-xxx XXXXXX

Listing. 2 Laboratory data evaluation. Complete blood count. Listing

| Centre-Patient | Sex | Age (years) | Visit | Treatment group | Test date | Parameter | Value | Measurement<br>units | H/N/L/ND | Significance<br>of the<br>deviation |
|---|---|---|---|---|---|---|---|---|---|---|
| xx-xxxx | XXXXX | xx.x | xxxxxxx | xxxxxxxxx | xxxx-xx-xx | xx.x | g/dL | N | xx.x | Clinically insignificant |
| xx-xxxx | XXXXX | xx.x | xxxxxxx | xxxxxxxxx | XXXX-XX-XX | XX.X | g/dL | N | xx.x | Clinically<br>significant |

Listing. 3 Laboratory data evaluation. Blood biochemistry. Listing Same as Listing 2

Listing. 4 Laboratory data evaluation. Urinalysis. Listing Same as Listing 2